CLINICAL TRIAL: NCT02220374
Title: Supportive Tape for Arthritis of the Proximal Interphalangeal Joint: A Two Group Parallel Randomised Placebo Controlled Trial
Brief Title: A RCT of Supportive Finger Tape for PIPJ Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mid Yorkshire Teaching NHS Trust (Other)
Responsible Party: Principal Investigator, Ryckie Wade, Core Surgical Trainee, Mid Yorkshire Teaching NHS Trust
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 14/YH/1040
Record Dates: First submitted 2014-08-16; First posted 2014-08-19 (Estimated); Last update posted 2017-08-31 (Actual); Status verified 2017-08

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis; Finger; Supportive; Tape; Pain; Function; Trial
MeSH Terms: conditions — Osteoarthritis; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Supportive Finger Tape (Experimental): Participants will be randomised to either placebo or supportive taping
  Interventions: Other: Supportive Finger Tape

INTERVENTIONS:
Other: Supportive Finger Tape — Dorsally applied elasticated tape may or may not improve the kinetics of the PIPJ and therefore reduce pain as well as improve function

SUMMARY:
Oesteoarthritis of the joints of the finger(s) is a common problem. The first-line treatment involves pain killers taken either as tablets, gels, or patches. Secondly, some joints are amenable to injections of steroids and anaesthetic agents. Finally, as a last resort, some joints may be fused or replaced with prosthetic joints by Hand Surgeons. We are investigating whether supportive taping of the painful finger joint reduces pain and improves function, and whether this treatment could be used to substitute pain killers, injections or surgery. We hypothesise that supportive finger tape may improve pain, improve the stability of the joint and thereby improve day-to-day hand function too. We will investigate this through a two-group parallel randomised controlled trial whereby one group will receive the treatment taping and the other group will receive a theoretically placebo taping configuration. We will measure pain daily, hand function and adverse events.

DETAILED DESCRIPTION:
Introduction:

Osteoarthritis (OA) of the interphalangeal joints of the hand is the most common age-related joint disorder worldwide, affecting the hand(s) of up to 67% of the elderly population. At least 18.2% of such patients have OA of at least one proximal interphalangeal joint involved and it is the second leading cause of hand pain after osteoarthritis of the thumb carpometacarpal joint. In the UK, 3% of the population seek medical attention for the symptoms of their hand arthritis, with the main complaints being pain, reduced grip strength, functional limitations with day-today activities (eg. dressing, eating and drinking, taking medication, writing, etc), stiffness and deformity.

Currently, the treatment of osteoarthritis of the finger joints is limited to four different avenues which carry their own limitation(s) and potential complications. Firstly, conservative measures such as physiotherapy with or without splints and compression garments, alterations in the execution of daily activities and avoidance of environmental triggers (eg. cold and wet weather) - these carry substantial time commitments and interference with normal life. Secondly, analgesics either by the oral, transcutaneous or topical routes may be used - these medication may cause drowsiness, confusion, constipation, collapse, kidney injury, stomach ulcers and bleeding, as well as other undesirable effects which may in-turn precipitate life-threatening illnesses. Thirdly, joints may be injected with steroids and anaesthetic agents which is both diagnostic and therapeutic - however, this too carries risks of septic arthritis, tendon attrition and paradoxical exacerbation of symptoms. Finally, surgery may be offered to either replace the joint with a prosthesis or fuse it with metal screw(s) and wire(s) - surgery carries significant risk of infection and damage to vessels or nerves, which may render the finger useless or even lead to amputation.

With the current available treatments carrying significant limitations, we have conceptualised a treatment which confers minimal (no proven) risk and may be of benefit to some individuals based on a current theorised treatment of supportive taping. The Kinesio® taping system is a well-known product used by many athletes to support their joints and improve performance. The elasticated latex tape is applied to the skin overlying a joint, in a specific orientation in order to provide theoretical benefits including: physical support for misaligned joints, increased recoil of the joint back to the anatomical position, and reduce swelling by improving lymphatic flow. A recent systematic review concluded that the most significant benefit from Kinesio® taping was reduced pain in large joints (eg. shoulder, knee and ankle). The reason for this is not well understood but may be related to stimulation of cutaneous and peri-articular mechanoreceptors, physically re-aligned/support of the joint surface or a placebo effect.

At present, the Kinesio® system is not ideal for patients with finger joint osteoarthritis for two reasons - there is no commercially available tape which is small enough to apply to the finger and the latex component may prevent some patients from using it. However, a latex free substitute is readily available in the hospital setting, which has similar properties (ie. adhesive and elasticated) which is safe and cheaper - Suture Strips® by Derma Sciences™.

Research on normal healthy subjects has shown that supportive taping of fingers improves perceived grip strength. Further, in patients with injured fingers, supportive taping increases actual grip strength in particular positions/actions. We know that patients with painful thumb joints benefit from supportive taping as it improves their joint alignment and therefore function. However, to-date there have been no studies on the role of finger PIPIJ taping to reduce the pain of arthritis. We hypothesise that by transferring the proven benefits of supportive taping on other bodily regions (ie. pain reduction, improved joint alignment, mechanical support as well as other undefined benefits) that patients may benefit from supportive taping of the PIPJ of the finger.

Rationale:

The current treatment modalities for finger joint arthritis carry significant risk of undesirable and potentially dangerous complications. We propose a simple method of supportive taping which may improve patient's pain and function, within conferring the risk of adverse events.

Aims:

We aim to investigate the effectiveness of supportive tape on the perceived pain of PIPJ osteoarthritis in a single digit of one hand. We also aim to investigate its impact on hand function and will undertake an economic analysis in comparison to current available treatments.

Type of study:

A pragmatic blocked two-group parallel randomised placebo controlled trial.

Research questions:

Primary research question;

1. Does supportive taping of the PIPJ of the finger effect perceived pain

Secondary research questions:

1. Does supportive taping of the PIPJ of the finger effect functional capability
2. Does supportive taping of the PIPJ of the finger effect have any significant adverse or undesirable effects
3. Does supportive taping of the PIPJ of the finger effect represent and economically feasible alternative to other current therapies
4. Does placebo taping of the PIPJ of the finger effect patient reported pain
5. Does placebo taping of the PIPJ of the finger effect objective hand function

ELIGIBILITY:
Inclusion criteria:

All adult patients (≥18 years old) with chronic osteoarthritis of the PIPJ of any finger.

Exclusion criteria:

Patients meeting any of the below criteria will be excluded:

* Patients lacking capacity to consent (unable to understand, retain, weigh up or communicate their decision)
* Patients (and/or their carers) who lack the dexterity to cut and apply the Suture Strips to the painful finger.
* Patients with active infection or unhealed wounds on the same hand as this may confound the level of pain experienced.
* Dermatological conditions or vulnerable dorsal finger skin on the proposed trial finger, which may be exacerbated or damaged respectively by the applicable/removal of tape

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2014-11; Primary Completion 2016-06-01 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
Change in Pain | 1 week
  We will measure the change in pain in the trial PIPJ by comparing reported pain without supportive tape over 7 days, to the reported pain over 7 days with supportive tape applied to the finger

SECONDARY OUTCOMES:
Hand Function | 3 weeks
  Using the Quick-DASH and qualitative means, we will capture whether supportive finger tape affects daily activities and hand function.
Adverse outcomes | 3 weeks
  We will investigate (through quantitative and qualitative means) whether this supportive finger tape caused any adverse events, such as rashes, skin tears or otherwise.

OTHER OUTCOMES:
Economic impact | 3 weeks
  We will speculate and compare the costs of supportive finger tape with other treatments, suggesting its economic feasibility

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Southern, MBBS FRCS(Plast), Study Director — Pinderfields General Hospital, Wakefield
Locations (1):
- Pinderfields General Hospital, Wakefield, United Kingdom